CLINICAL TRIAL: NCT03821675
Title: Electrical Stimulation as an Adjunctive Therapy to Accelerate Wound Healing in People With Diabetic Foot Ulcers - A Randomized Controlled Trial
Brief Title: Electrical Stimulation to Accelerate Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Avazzia, Inc (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-44704
Record Dates: First submitted 2019-01-24; First posted 2019-01-30 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Diabetes; Diabetic Foot Ulcer; Peripheral Neuropathy; Peripheral Arterial Disease
Keywords: electrical stimulation; wound healing; skin perfusion; home based therapy; diabetic foot; Foot ulcer
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Peripheral Nervous System Diseases; Peripheral Arterial Disease; Foot Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Devices may be active or sham.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Electrical Stimulation - Active (Active Comparator): Subjects will receive an active electrical stimulation device to wear for 1 hour daily for 4 weeks.
  Interventions: Device: Electrical Stimulation - Active
- Electrical Stimulation - Sham (Sham Comparator): Subjects will receive a sham electrical stimulation device to wear for 1 hour daily for 4 weeks.
  Interventions: Device: Electrical Stimulation - Sham

INTERVENTIONS:
Device: Electrical Stimulation - Active — Subjects will receive an active electrical stimulation device to wear for 1 hour daily for 4 weeks.
  Arms: Electrical Stimulation - Active
Device: Electrical Stimulation - Sham — Subjects will receive a sham electrical stimulation device to wear for 1 hour daily for 4 weeks.
  Arms: Electrical Stimulation - Sham

SUMMARY:
A clinical study at the Baylor College of Medicine, Division of Vascular Surgery and Endovascular Therapy, is being proposed to test the efficacy of a novel electrical stimulation platform named the Tennant Biomodulator designed by AVAZZIA to accelerate wound healing, relieve pain and improve mobility in patients with diabetic foot ulcers.

DETAILED DESCRIPTION:
Electrical stimulation may offer a unique treatment option to heal complicated and recalcitrant wounds, improve flap and graft survival, and even reduce the likelihood of ulceration. Electrical stimulation has been suggested to reduce infection, improve cellular immunity, increase perfusion, relieve pain, improve plantar sensation, and accelerate wound healing.

Electrical stimulation could have positive effect on not only increasing skin perfusion in patients with diabetes but also could improve mobility and balance via enhancing plantar sensation as demonstrated in our recent study. Thus, plantar stimulation not only may be beneficial to accelerate wound healing in diabetic foot ulcer (DFU) patients but also may assist to improve mobility and reduce the likelihood of recurrence of ulcers.

This study is proposed to examine the effectiveness of an innovative portable electrical stimulation platform (Tennant Biomodulator by AVAZZIA) to accelerate wound healing in DFU patients. It is hypothesized that 1) electrical stimulation will have an immediate effect on increasing skin perfusion (immediate benefit) and 2) daily use of the Tennant Biomodulator for 4 consecutive weeks is effective to speed up wound healing, increase skin perfusion, reduce pain, and improve balance and mobility in DFU patients (long term benefit)

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* 18-85 years old
* Clinically confirmed diabetes (ADA criteria)
* Clinically confirmed Peripheral Neuropathy
* One or more active non-infected ulcers
* Subject or responsible caregiver is willing and to maintain the required offloading (as applicable the location of the ulcer) and applicable dressing changes and electrical stimulation application.

Exclusion Criteria:

* Subject has a demand-type cardiac pacemaker, implanted defibrillator or other implanted electronic device
* Is pregnant
* Is nursing or actively lactating
* Has Renal Disease
* Active wound infection
* Active Charcot foot
* Non-ambulatory (unable to walk 40 feet with or without assistive device)
* Bilateral AK/BK amputation
* Active drug/alcohol abuse
* Dementia or impaired cognitive function
* Excessive lymphedema
* Osteomyelitis and/or gangrene
* Unable to comply with research appointments (e.g. long travel) Wide spread malignancy or systemically imumno-compromising disease
* Subject has a history of or any intercurrent illnesses or conditions that would compromise the safety of the subject according to judgement of a qualified wound specialist.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active: Subjects will receive an active electrical stimulation device to wear for 1 hour daily for 4 weeks.
- Sham: Subjects will receive a sham electrical stimulation device to wear for 1 hour daily for 4 weeks.
Period: Overall Study
Arm/Group | Active | Sham
Started | 19 | 19
Completed | 16 | 17
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Sham | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (13.8) | 61.4 (11.2) | 63.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Skin Perfusion in Response to Electrical Stimulation Therapy
Description: Lower-extremity skin perfusion will be assessed using a skin perfusion pressure device (PADIQ Sensilase). This device emerges pressure with a cuff placed around the calf muscle that has internal sensors. Then, the cuff is slowly released letting circulation to re-enter which is detected by the sensors.
Time Frame: Change at 4 weeks from baseline.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Active | Sham
Number analyzed (Participants) | 16 | 17
mmHg | 65.1 (19.1) | 72.2 (18.1)

2. Primary Outcome: Change in Wound Size in Response to Electrical Stimulation Therapy
Description: Wound size will be assessed with a Sillouette Star 3D Camera that detects width, length, and depth of wounds that automatically gives you a cm2 area.
Time Frame: Change at 4 weeks from baseline
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Active | Sham
Number analyzed (Participants) | 16 | 17
cm2 | 5.8 (8) | 3.2 (8.7)

3. Secondary Outcome: Change in Plantar Sensation in Response to Electrical Stimulation
Description: change in plantar sensation will be assessed with a vibration pressure threshold device placed on the heel.
Time Frame: Change at 4 weeks from baseline.
Measure: Mean (Standard Deviation); unit: Volts
Arm/Group | Active | Sham
Number analyzed (Participants) | 16 | 17
Volts | 20.2 (14) | 32.1 (9.2)

4. Secondary Outcome: Change From Baseline to 60 Minutes in Tissue Oxygen Saturation in Response to Electrical Stimulation
Description: Plantar tissue oxygen saturation will be assessed with Near infrared Spectroscopy device (KENT Imaging) at 60 minutes from baseline.
Time Frame: Change at 60 minutes from baseline.
Population: Active electrical stimulation was performed during one hour on all participants before randomization.
Measure: Mean (Standard Deviation); unit: SatO2%
Groups:
- Active: Subjects will receive an active electrical stimulation device to wear for 1 hour
- Sham: Subjects did not receive sham device for this outcome measure.
Arm/Group | Active | Sham
Number analyzed (Participants) | 38 | 0
SatO2% | 73.5 (12.5) |

5. Secondary Outcome: Change in Tissue Oxygen Saturation in Response to Electrical Stimulation
Description: Plantar tissue oxygen saturation will be assessed with Near infrared Spectroscopy device (KENT Imaging)
Time Frame: Change at 4 weeks from baseline.
Measure: Mean (Standard Deviation); unit: SatO2%
Arm/Group | Active | Sham
Number analyzed (Participants) | 16 | 17
SatO2% | 72.3 (21.5) | 73.9 (12.1)

6. Other Pre Specified Outcome: Change From Baseline in Skin Perfusion in Response to Electrical Stimulation
Description: as for outcome 1
Time Frame: an average of 60 minutes from baseline
Population: Active electrical stimulation was performed during one hour on all participants before randomization.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Active | Sham
Number analyzed (Participants) | 38 | 0
mmHg | 79.9 (18.3) |

ADVERSE EVENTS:
Time Frame: an average of 4 weeks from baseline.
Description: 0
Groups:
- Active: intervention
- Sham: control
Arm/Group | Active | Sham
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT03821675/Prot_005.pdf
  • Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT03821675/SAP_004.pdf